CLINICAL TRIAL: NCT06281990
Title: The Effect of Pre-admission Education Given to Bariatric Surgery Patients on Postoperative Recovery
Brief Title: Education and Information for Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, pinar ongun, Assistant Professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BAUN-SBF-PO-01
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgeries; Education of Patients
Keywords: patient education; bariatric surgery; laparoscopic sleeve gastrectomy
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: There are two groups in the research: control and intervention groups.
Who Masked: Care Provider, Investigator
Masking Description: The researcher (YY) provided education in the outpatient clinic. The nurses and surgical team members working in the surgical ward were blinded (FÇ in the research group was blinded).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group received standard care.
- Intervention group (Experimental): 1:Patients who were planned to undergo sleeve gastrectomy surgery were informed about the perioperative period when they came to the outpatient clinic2-4weeks before surgery and were educated about the exercises to be performed before and after surgery. The content of this education included pain management, breathing exercises,foot rotation, and leg exercises. In addition, the education book prepared by the researchers was given to the patients to make the education and information permanent until the day of surgery.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — 1. Patients who were planned to undergo sleeve gastrectomy surgery were informed about the perioperative period when they came to the outpatient clinic2-4weeks before surgery and were educated about the exercises to be performed before and after surgery. The content of this education included pain management, breathing exercises,foot rotation, and leg exercises. In addition, the education book prepared by the researchers was given to the patients to make the education and information permanent until the day of surgery.
  2. When the patient was hospitalized, anxiety level with the Trait Anxiety scale and pain level with VAS were determined one day before surgery.
  3. Postoperatively, the patient's pain level before analgesics every 4-6hours for 2days, the patient's anxiety level with the State Anxiety Scale one day after surgery, the development of complications in the postoperative period, vital signs were evaluated, and the duration of hospitalization was recorded.
  Arms: Intervention group

SUMMARY:
The study aimed to investigate the effect of pre-admission education given to bariatric surgery (laparoscopic sleeve gastrectomy) patients on preoperative and postoperative anxiety, postoperative pain, and patient vital signs.

DETAILED DESCRIPTION:
Aim: The study aimed to investigate the effect of pre-admission education given to laparoscopic sleeve gastrectomy patients on preoperative and postoperative anxiety, postoperative pain, and patient vital signs.

Materials and Methods: This randomized, controlled, experimental, single-blinded study was conducted with 68 patients who met the inclusion criteria and underwent laparoscopic sleeve gastrectomy in the general surgery clinic of a university hospital between December 2022 and October 2023. The CONSORT checklist was used as a guide. Data were collected using the "Perioperative Form," "Visual Analog Scale, and "State-Trait Anxiety Scale" All patients were operated on by the same physicians and received standard perioperative care. Intervention group patients were informed and educated about the surgical process in the outpatient clinic. Anxiety levels were determined one day before surgery. In the postoperative period, vital signs, anxiety, and pain levels were measured 8 times during 48 hours.

Stage 1: Patients who were planned to undergo sleeve gastrectomy surgery were informed about the perioperative period in an appropriate room when they came to the outpatient clinic 2-4 weeks before surgery and were educated about the exercises to be performed before and after surgery. The content of this education included pain management, breathing exercises (use of trifle, deep breathing, coughing), foot rotation, and leg exercises. In addition, the education book prepared by the researchers was given to the patients to make the education and information permanent until the day of surgery.

Stage 2: When the patient was hospitalized, anxiety level with the Trait Anxiety Scale and pain level with VAS were determined one day before surgery.

Stage 3: Postoperatively, the patient's pain level before analgesics every 4-6 hours for 2 days, the patient's anxiety level with the State Anxiety Scale one day after surgery, the development of complications in the postoperative period, vital signs were evaluated, and the duration of hospitalization was recorded

ELIGIBILITY:
Inclusion Criteria:

* being conscious
* not having a diagnosis of psychiatric disease,
* being 18 years of age or older,
* undergoing their first bariatric surgery,

Exclusion Criteria:

* not being conscious
* Having a diagnosis of psychiatric disease,
* Being 18 years of age or younger,
* Not having bariatric surgery for the first time
* to be reoperated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Data collection form | preoperative phase
  It consists of a total of 25 questions, including questions such as age, gender, educational status, previous surgery, counseling and training status, duration of surgery, and postoperative complications, vital sigs
Visual Analog Scale (VAS) | Pain level with VAS were determined one day before surgery; postoperatively, the patient's pain level before analgesics every 4-6 hours for 2 days
  Pain assessment was performed with VAS. "0" indicates no pain, and "10" indicates the most severe unbearable pain.
State-Trait Anxiety Inventory (STAI) | Anxiety level with STAI were determined one day before surgery; postoperatively, the patient's anxiety level with the STAI scale one day after surgery
  The inventory measures state and trait anxiety levels in normal and abnormal individuals. Turkish validity-reliability study was conducted. The STAI consists of two scales of twenty items each, measuring state and trait anxiety levels. The "STAI FORM" questionnaire form of the STAI scale used to measure the state anxiety of patients will be used in the study. The State Anxiety Scale determines how an individual feels at a given moment and under certain conditions. Trait Anxiety Inventory is a measurement tool consisting of statements that indicate how a person usually feels. In answering the State-Trait Anxiety Scale, one is asked to select and mark one of the options "not at all, a little, a lot, completely" according to the severity of the feelings, thoughts, or behaviors expressed by the items. Responses range from 1 to 4. A high score indicates a high level of anxiety. A high score indicates a "high anxiety" level, and a low score indicates a "low anxiety" level.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Ongün, Principal Investigator — Balıkesir Üniversitesi; Sibel Karaca Sivrikaya, Principal Investigator — Balıkesir Üniversitesi
Locations (1):
- Pınar Ongün, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share the data whenever requested if it will be used in research such as meta-analysis.